CLINICAL TRIAL: NCT02959931
Title: Postprandial Physiological Effects of a High Potassium Meal in Patients With Hypertension
Brief Title: Postprandial Effects of a High Potassium Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MSH 13-0088-A
Record Dates: First submitted 2015-12-22; First posted 2016-11-09 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Hypertension
Keywords: Dietary Potassium
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High potassium meal (Experimental): In this arm individuals will be provided with a breakfast meal that provides ~2400 mg of dietary potassium.
  Interventions: Other: High Potassium Meal
- Low potassium meal (Active Comparator): In this arm individuals will be provided with a breakfast meal that provides ~540 mg of dietary potassium.
  Interventions: Other: Low Potassium Meal

INTERVENTIONS:
Other: High Potassium Meal — Breakfast meal that provides ~2400 mg of dietary potassium. Meals are isocaloric.
  Arms: High potassium meal
Other: Low Potassium Meal — Breakfast meal that provides ~540 mg of potassium. Meals are isocaloric.
  Arms: Low potassium meal

SUMMARY:
The investigators aim to evaluate the acute effects of potassium supplementation achieved by ingestion of potassium rich food, on vascular health.

DETAILED DESCRIPTION:
Many studies have shown that an increase in potassium through the diet or through potassium pills helps to lower blood pressure. Also, the amount of oral potassium taken can improve how well the participants blood vessels work. These studies have focused on potassium given in the form of a pill. The investigators are interested in the effect of potassium consumed through food sources and how it will effect arterial health and blood pressure. The world health organization (WHO) recommends a K⁺ intake of at least 3510 mg/day from food for adults, excluding those with impaired K⁺ excretion. In this study the investigators aim to provide approximately 75% (approximately 2000 mg) of the total daily recommended intake for potassium in one meal. The investigators do not know whether dietary potassium (not pill form) will acutely improve the arterial health and if it will cause a decrease in blood pressure. The investigators hypothesis to see an improvement in vascular function following a high potassium meal compared to a low potassium meal.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years
* Normal sinus rhythm
* A diagnosis of hypertension on medical therapy with an ambulatory systolic blood pressure <160 mmHg and diastolic blood pressure <90 mmHg, or a diagnosis of stable coronary artery disease

Exclusion Criteria:

* Recent hospital admission due to an cardiovascular events
* Serum K+ concentration >5.0 mmol/L
* Current smoking
* Women who are pregnant
* Diabetic patients - patients receiving insulin therapy
* Glomerular filtration rate < 90mls/min/1.73m2
* On loop diuretic therapy
* Food allergies and/or intolerance to meal items

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Flow Mediated Dilatation | Flow Mediated Dilatation will be assessed over 2 clinic visits, at 3 times points with in each visit; pre-prandial and post-prandial at 60 min and 120 min
  Flow Mediated Dilatation is a method used to measure endothelial-dependent regulation of conduit artery tone(Joannides R, 1995).

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No